CLINICAL TRIAL: NCT07210437
Title: Longitudinal Autonomic Characterization as a Predictor for Secondary Medical Complications Post-SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Ryan J. Solinsky, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-003333
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Spinal Cord Injury (Experimental)
  Interventions: Diagnostic Test: Tests of sympathetic inhibition; Diagnostic Test: Tests of above level sympathetic activation; Diagnostic Test: Testing of below level sympathetic activation
- Acute Spinal Cord Injury (Experimental)
  Interventions: Diagnostic Test: Tests of sympathetic inhibition; Diagnostic Test: Tests of above level sympathetic activation; Diagnostic Test: Testing of below level sympathetic activation

INTERVENTIONS:
Diagnostic Test: Tests of sympathetic inhibition — Bolus phenylephrine infusion using the Oxford technique will generate the need to inhibit sympathetic activity. Similarly, resting state Mayer waves will be assessed with regard to heart rate and blood pressure responses.
Diagnostic Test: Tests of above level sympathetic activation — Cold pressor test of the hand will be used to cause sympathetic activation. Valsalva's maneuver will assess the ability to buffer against blood pressure fall (phase II).
Diagnostic Test: Testing of below level sympathetic activation — Cold pressor test of the foot and bladder pressor response will be tested.

SUMMARY:
The purpose of this research is to learn about how the body is able to balance changes in blood pressure, how that changes over time, and how these changes impact a participant's risk of developing medical problems.

ELIGIBILITY:
Inclusion criteria

* 18-75 years old
* Spinal cord injury with neurological level of injury from C6-T12
* ASIA Impairment Scale A-D.
* Either acute SCI <3 months prior (n=10) or chronic SCI (>1 year since injury, n=8).

Exclusion criteria

* Symptoms of cardiovascular (including, but not limited to: hypertension, stroke, chest pain, etc.), respiratory, peripheral neurological or autonomic disease (particularly diabetes mellitus requiring treatment);
* Women who are pregnant or lactating
* Taking or being administered a medication known to potentially have adverse interactions with phenylephrine
* In the judgement of the principal investigator, any illness or condition that will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Valsalva Maneuver Phase II | During laboratory diagnostic testing session
  Presence or absence of phase II on Valsalva maneuver testing, which takes approximately 15 seconds to complete. This will be repeated x3.

SECONDARY OUTCOMES:
Beat-to-beat heart rate | During laboratory diagnostic testing session
  Electrocardiogram will record continuous measures with changes in R-R interval (ms) quantified and compared to baseline.
Beat-to-beat blood pressure | During laboratory diagnostic testing session
  Non-invasive continuous blood pressure monitors will be used, with changes in systolic and diastolic pressure (in mmHg) from resting baseline measured.
Continuous galvanic skin response | During laboratory diagnostic testing session
  Changes from resting state conductance with be quantified with a smartwatch.
Quantify autonomic dysreflexia and orthostatic hypotension | Baseline, prior to laboratory diagnostic testing session
  Participants will be given the Autonomic Dysfunction Following Spinal Cord Injury questionnaire (score range 0-436, with higher scores indicating more autonomic dysfunction).
Respiration | During laboratory diagnostic testing session
  Elastic respiratory transducer bands around mid-chest and upper abdomen will monitor breathing depth and frequency.
Beat-by-Beat Popliteal and Brachial Blood Flow | During laboratory diagnostic testing session
  The investigators will use Doppler derived flow velocities to estimate whole limb blood flow through the popliteal and brachial arteries
Immunology Blood Draw | During laboratory diagnostic testing session
  Baseline samples will be collected and compared against changes to blood pressure.
Serum Catecholamines and Cortisol | During laboratory diagnostic testing session
  Baseline resting catecholamines (norepinephrine, epinephrine, dopamine) and cortisol will be drawn from the IV after 10 minutes of quiet rest at baseline and prior to bladder filling or foot cold pressor. Just prior to the conclusion of this testing, an additional blood draw will take place through the IV to assess changes in these levels.
Pressure-induced vasodilation | During laboratory diagnostic testing session
  Changes to skin blood flow following a gradual change in pressure to the skin surface area. Laser doppler will be used to monitor changes in blood flow.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Solinsky, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Solinsky R, Burns K, Hamner JW, Singer W, Taylor JA. Characterizing preserved autonomic regulation following spinal cord injury: Methods of a novel concerted testing battery and illustrative examples of a new translationally focused data representation. medRxiv [Preprint]. 2024 Jun 1:2024.05.31.24308290. doi: 10.1101/2024.05.31.24308290. PMID 38854077